CLINICAL TRIAL: NCT04344028
Title: Examining the Potential for Placebo Effects in Cognitive Training
Brief Title: Examining the Effectiveness of Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of California, Riverside (Other); University of California, Irvine (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019-1378; 1R56AG063952-01 (NIH); A487400 (Other: UW Madison); L&S/PSYCHOLOGY (Other: UW Madison)
Record Dates: First submitted 2020-04-07; First posted 2020-04-14 (Actual); Results first posted 2022-10-20 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2022-10

CONDITIONS: Cognitive Change
Keywords: Cognitive Training

STUDY DESIGN:
Intervention Model Description: The design is a 2 (positive expectations/negative expectations) x 2 (true cognitive training intervention x control cognitive training intervention) randomized controlled trial.
Who Masked: Participant, Investigator
Masking Description: Researchers and participants will be blind to the conditions assigned to the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- True Cognitive Training Placebo (Experimental): Participants will receive a positive expectation message (e.g., "Previous research has shown that training with this program improves performance on other tasks.") and will complete approximately 7 hours of a cognitive training program that has previously been shown to improve cognition.
  Interventions: Behavioral: True Cognitive Training Program; Behavioral: Positive Expectation Induction
- True Cognitive Training Nocebo (Active Comparator): Participants will receive a negative expectation message (e.g., "Previous research has shown that training with this program decreases performance on other tasks.") and will complete approximately 7 hours of a cognitive training program that has previously been shown to improve cognition.
  Interventions: Behavioral: True Cognitive Training Program; Behavioral: Negative Expectation Induction
- Control Cognitive Training Placebo (Placebo Comparator): Participants will receive a positive expectation message (e.g., "Previous research has shown that training with this program increases performance on other tasks.") and will complete approximately 7 hours of control training program that has not previously been shown to improve cognition.
  Interventions: Behavioral: Control Cognitive Training Program; Behavioral: Positive Expectation Induction
- Control Cognitive Training Nocebo (Sham Comparator): Participants will receive a negative expectation message (e.g., "Previous research has shown that training with this program decreases performance on other tasks.") and will complete approximately 7 hours of control training program that has not previously been shown to improve cognition.
  Interventions: Behavioral: Control Cognitive Training Program; Behavioral: Negative Expectation Induction

INTERVENTIONS:
Behavioral: True Cognitive Training Program — The training program is a personal device-based adaptive version of a visual N-back task.
  Arms: True Cognitive Training Nocebo; True Cognitive Training Placebo
Behavioral: Control Cognitive Training Program — The training program is a personal device-based adaptive version of a knowledge task (control).
  Arms: Control Cognitive Training Nocebo; Control Cognitive Training Placebo
Behavioral: Positive Expectation Induction — The message given to the participants emphasizes that the given training results in a positive change in cognitive abilities.
  Arms: Control Cognitive Training Placebo; True Cognitive Training Placebo
Behavioral: Negative Expectation Induction — The message given to the participants emphasizes that the given training results in a negative change in cognitive abilities.
  Arms: Control Cognitive Training Nocebo; True Cognitive Training Nocebo

SUMMARY:
The present study addresses whether placebo effects can possibly account for previous findings in the field, as well as ascertains whether placebo-based mechanisms can be deliberately harnessed for impact. The design is a 2 (positive expectations/negative expectations) x 2 (true cognitive training intervention x control cognitive training intervention) Randomized Controlled Trial (RCT). Participants will be recruited from site-affiliated participant pools or email lists.

Participants will first undergo a pre-test battery where various cognitive abilities are assessed via computerized programs. They will also fill out various surveys about personality traits/internal dispositions that may predict the extent to which they are susceptible to placebo effects.

After pre-testing, participants will be randomized to an expectations group (positive/negative) and a training protocol (active/control). Participants are then given their group appropriate expectation script. In the positive expectations group, participants receive training described as having previous research supporting its use as a method to enhance cognitive abilities. In the negative expectations group, participants receive training described as having previous research suggesting that it is unlikely to change cognitive abilities or may even decrease cognitive abilities.

The participants will then be given instructions regarding how to do their training task. Participants will be asked to complete 10 sessions of training within 15 days. The active training will be a standard working memory (N-back) training task. The control training will be a trivia/quiz training task.

After they have completed 10 sessions, participants will complete a "mid-test" session to undergo a battery of perceptual/cognitive tasks. Participants will be told that the perceptual/cognitive tests are identical to those that they took at pre-test. However, in reality, for participants in the "positive expectations" groups, these will be altered to actually be easier than they were at pre-test. For participants in the "negative expectations" groups the tasks will be made more difficult.

Participants will then be asked to complete another set of 10 training sessions on their devices within 15 days before completing the post-test. The post-test will be identical to the pre-test. All participants will then be extensively debriefed (e.g., all deceptions will be made clear). On a separate day, participants will then complete a second post-test that is identical to the pre-test and first-post test.

DETAILED DESCRIPTION:
This study examines the extent to which working memory training may give rise to cognitive benefits and the extent to which these effects can be explained by, or augmented by, placebos.

It is predicted that:

1. Significant placebo effects will be found in cognitive training, both at the immediate post-test and the second post-test after participants were debriefed about the placebo effects.
2. Adaptive N-back training will produce larger gains than adaptive Knowledge training.

Participants will be assigned to either an online or in-person version of the study depending upon the guidelines for participant interactions that are in force at the time (if only one version is allowable under current guidelines participants will be assigned to the allowable version).

Pre-Test Cognitive Assessments: For each domain, two separate measures will be utilized to ensure that any observed results are not specific to a given tasks, but are more generally representative for the six cognitive domains below.

1. Working Memory: The two measures will be a non-trained version of the N-back task and the O-Span task. In the N-back task, participants view a series of letters and are asked to indicate whether the current letter is the same as the letter "N" items back. The N-back levels will vary between 1- and 4-back. In the O-Span task, participants alternate between completing simple math problems (e.g., 3+(2x2)) and viewing single letters. At the end of a given sequence, the participants are asked to recall all of the letters that they had seen in the correct order. The number of letters to be recalled will range between 3 and 7.
2. Cognitive Flexibility: The two measures will be a standard task-switching paradigm and countermanding task. In the task switching task, on each trial, participants view a letter and a digit. The location of the pair instructs the participants to either categorize the letter as a consonant or vowel or else categorize the digit as even or odd. Trials can be either "non-switch trials" - in which the participant is asked to perform the same task as on the previous trial - or "switch trials" - in which the participant is asked to perform the opposite task as on the previous trial. In the countermanding task, participants are presented with two types of stimuli (e.g., dogs or monkeys) on either the right or the left side of the screen and are required to tap on one of two buttons on either the same side as the stimulus (e.g., dog; congruent trials) or on the opposite side of the stimulus (e.g., monkey; incongruent trials).
3. Visual Selective Attention: The two measures will be the Useful Field of View (UFOV) task and the Attentional Network Test (ANT; executive control trials only). In the UFOV, participants are briefly presented with a display consisting of 24 items (3 on each of the four radial spokes and the four obliques; evenly spaced). One of the items is a target (a sheriff's badge), while the remaining items are distractors (open boxes). The participants' task is to indicate upon which of the 8 spokes the target appeared. In the ANT, on each trial participants view a center arrow that faces either left or right. The arrow can be flanked on either side by either response compatible arrows (i.e., arrows facing in the same direction as the center arrow) or response incompatible arrows (i.e., facing the other direction). The participants' task is to indicate the direction that the center arrow is pointing.
4. Spatial Cognition: The two measures will be a standard mental rotation test and paper folding test. In the mental rotation task, participants are shown two images side by side. The images are either identical, but with one rotated relative to the other, or else are mirror-reversed and rotated copies of one another. The participants' task is to indicate whether the two items are identical or are mirror-reversed copies. In the paper-folding task, the participant is shown a depiction of a piece of paper being folded various ways before a hole is punched in the paper. The participants' task is to indicate what the paper will look like when it is unfolded.
5. Fluid Intelligence: The two measures of fluid intelligence will be the Raven's Advanced Progressive Matrices and a new matrix task (UCMRT) developed and implemented by PIs Jaeggi and Seitz. In each test item, the participant is presented with a grid of elements with one of the elements missing and is asked to identify the missing element that completes the grid pattern.
6. Vocabulary (control): Vocabulary will be assessed using the Mill-Hill vocabulary and the Shipley Institute of Living scales. These require participants to select the appropriate synonym for a target word among several alternatives.

Pre-Test Individual Differences Surveys: At Pre-test, participants will complete a series of surveys to assess demographic variables (e.g., age, gender, race/ethnicity, SES) as well as other individual difference factors that may be predictive of placebo-responsiveness. These include: Big 5 Personality Traits, Work and Family Orientation Scale (WOFO), Grit, Behavioral Avoidance/Inhibition scales (BIS/BAS), theories of intelligence, Schutte Self-Report Emotional Intelligence Test, and Meta-Cognitive Skills Scale.

Training Conditions: Participants will be assigned to either an experimental training condition (N-back training, which previous research has shown is associated with enhancements in general cognitive function) or a control training condition (explicit knowledge training, which previous research has shown is not associated with enhancements in general cognitive function). The cognitive training task will be an adaptive version of a visual N-back task used previously. Participants will be presented with a series of objects and will be asked to indicate whether the current stimulus matches the one presented n positions back in the sequence. An active knowledge training task (control) will be used in which participants will be asked to answer Graduate Record Examination-type (GRE) general knowledge, vocabulary, and trivia questions selected from a pool of approximately 5,000 questions. For every question, participants are required to pick one of four answer alternatives presented below the question and after their response are given the correct answer.

Explicit Expectation Induction: Participants will be assigned to either positive or negative expectations induction, which will be delivered via a slideshow. All instructions and descriptions of the to-be-trained task in the Positive Expectations groups will be designed to maximize participant belief in the effectiveness of the given training in inducing positive change in cognitive abilities or minimize participant belief in the Negative Expectations groups.

Associative Learning Mid-Tests: For the associative learning mid-tests, the same basic cognitive tasks employed at Pre-test will be altered to either provide evidence to the participant of "improved cognitive performance" (positive associative learning) or "diminished cognitive performance" (negative associative learning).

1. Working Memory Mid-Test Associative Learning Manipulations:

   O-Span: In the O-Span Associative Learning Mid-Test, task difficulty will be manipulated by either lessening the difficulty of the interleaved math problems (e.g., by using problems that only contain small numbers) or increasing the difficulty of the interleaved math problems.
2. Cognitive Flexibility Mid-Test Associative Learning Manipulation:

   Task-switching: In the task-switching test, several factors make the test more difficult. First is the number of task switches - fewer switch trials results in overall better performance. Second are the digits themselves. For instance, in the high/low task, digits closer to 5 are responded to more slowly than digits further from 5. Thus, in the Task-Switching Associative Learning Mid-Tests, the switch rate will be reduced (easier) or increased (harder) relative to the true assessments, and the distribution of digits that are displayed will include a greater or lesser percentage of easier items.

   Countermanding: In the Countermanding test, difficulty is most strongly associated with the presence of incongruent trials as well as switch trials. Thus, the Countermanding Mid-Test will have decreased or increased proportions of incongruent and switch trials from 50% to 30%/70%, respectively.
3. Visual Selective Attention Mid-Test Associative Learning Manipulation:

   UFOV: In the case of the UFOV, the simplest method to decrease difficulty is to increase presentation duration. Thus, in the UFOV Associative Learning Mid-tests, the proportion of long presentation duration trials will be increased (easier) or decreased (more difficult).

   ANT: In the case of the ANT, the Associative Learning Mid-tests will be made easier by increasing the proportion of neutral trials or made more difficult by decreasing the proportion of neutral trials and increasing the proportion of incompatible (most difficult) trials.
4. Spatial Cognition Mid-Test Associative Learning Manipulation:

   Mental Rotation: Difficulty in mental rotation is monotonically related to the degree of rotation between the two items (larger rotations = more difficult). The Mental Rotation Associative Learning Mid-tests will thus be constructed to contain a disproportionate number of items with either small (easier) or large (more difficult) orientation differences.

   Paper Folding: In the paper folding task, more difficult trials involve not only more total folds, but more partial folds and more angled partial folds. The Paper Folding Associative Learning Mid-tests will thus contain a disproportionate number of low total folds/low partial folds trials (easier) or high total folds/high partial folds trials (more difficult).
5. Fluid Intelligence Mid-Test Associative Learning Manipulation: All matrix items that will be utilized have a known level of difficulty. Thus, the Fluid Intelligence Associative Learning Mid-test sets will be created by mixing in a disproportionate number of easier/more difficult items for both Raven's and new matrix task created by PIs Seitz and Jaeggi.
6. Vocabulary Mid-Test Associative Learning Manipulation: As with the fluid intelligence test, the items have known levels of difficulty, and thus, the Associative Learning Mid-test will have a disproportionate number of easier/more difficult items for both the Mill-Hill vocabulary and the Shipley Institute of Living scales.

Knowledge of the Hypothesis Scales: Prior to Post-Test1, participants will be given two measures - the Perceived Awareness of the Research Hypothesis scale and the Expectation Assessment scale. Both measures are designed to assess the extent to which participants have internalized/believed the expectations that were meant to be induced.

Unblinding: Participants in all groups will be given a thorough debriefing after Post-Test1 and before Post-Test2 as to the goals of the study, the conditions, and any deception that they may have been subject to.

Post-Test1 and 2 will be identical to the Pre-test cognitive tests (new trials/items will be used in all cases).

ELIGIBILITY:
Inclusion Criteria:

* Self-reported normal or corrected-to-normal vision
* No known neurological impairments (this includes any neurological impairments that would negatively impact participants' ability to perform perceptual or cognitive tasks or to complete long-term cognitive training; this could include neurological damage due to stroke in various brain areas; seizure conditions that would preclude the ability to view flashing images; motor control issues that preclude the ability to respond via button presses; etc.).
* Access to the internet, a computer, and a hand-held device, such as a cell phone or tablet (online version only)

Exclusion Criteria:

* Self-reported non-normal or non-corrected-to-normal vision
* Neurological impairments
* No access to the internet, a computer, or a hand-held device (online version only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Seitz, PhD, Principal Investigator — University of California, Riverside; Susanne Jaeggi, PhD, Principal Investigator — University of California, Irvine
Locations (3):
- United States (3):
  - University of California, Irvine, Irvine, California
  - University of California, Riverside, Riverside, California
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (anonymized).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available persistently at the conclusion of the study.
Access Criteria: There are no access criteria.

REFERENCES:
- [Background] Jaeggi SM, Studer-Luethi B, Buschkuehl M, Su Y, Jonides J, Perrig WJ. The relationship between n-back performance and matrix reasoning - implications for training and transfer. Intelligence. 2010; 38: 625-635.
- [Background] Jaeggi SM, Buschkuehl M, Jonides J, Shah P. Short- and long-term benefits of cognitive training. Proc Natl Acad Sci U S A. 2011 Jun 21;108(25):10081-6. doi: 10.1073/pnas.1103228108. Epub 2011 Jun 13. PMID 21670271
- [Background] Conway AR, Kane MJ, Engle RW. Working memory capacity and its relation to general intelligence. Trends Cogn Sci. 2003 Dec;7(12):547-52. doi: 10.1016/j.tics.2003.10.005. PMID 14643371
- [Background] Unsworth N, Heitz RP, Schrock JC, Engle RW. An automated version of the operation span task. Behav Res Methods. 2005 Aug;37(3):498-505. doi: 10.3758/bf03192720. PMID 16405146
- [Background] Strobach T, Frensch PA, Schubert T. Video game practice optimizes executive control skills in dual-task and task switching situations. Acta Psychol (Amst). 2012 May;140(1):13-24. doi: 10.1016/j.actpsy.2012.02.001. Epub 2012 Mar 14. PMID 22426427
- [Background] Davidson MC, Amso D, Anderson LC, Diamond A. Development of cognitive control and executive functions from 4 to 13 years: evidence from manipulations of memory, inhibition, and task switching. Neuropsychologia. 2006;44(11):2037-78. doi: 10.1016/j.neuropsychologia.2006.02.006. Epub 2006 Mar 31. PMID 16580701
- [Background] Ball KK, Beard BL, Roenker DL, Miller RL, Griggs DS. Age and visual search: expanding the useful field of view. J Opt Soc Am A. 1988 Dec;5(12):2210-9. doi: 10.1364/josaa.5.002210. PMID 3230491
- [Background] Fan J, McCandliss BD, Sommer T, Raz A, Posner MI. Testing the efficiency and independence of attentional networks. J Cogn Neurosci. 2002 Apr 1;14(3):340-7. doi: 10.1162/089892902317361886. PMID 11970796
- [Background] Cooper L, Shepard R Chronometric studies of the rotation of mental images. In Visual Information Processing, W. Chase, ed. (New York, NY: Academic Press). 1973; 135-142.
- [Background] Lovett A, Forbus K. Modeling Spatial Ability in Mental Rotation and Paper-Folding. Proceedings of the 35th Annual Meeting of the Cognitive Science Society. 2013
- [Background] Raven JC, Court JH, Raven J. Manual for Raven's progressive matrices and vocabulary scales: Advanced Progressive Matrices Sets I and H. London: H. K. Lewis. 1983
- [Background] Pahor A, Stavropoulos T, Jaeggi SM, Seitz AR. Validation of a matrix reasoning task for mobile devices. Behav Res Methods. 2019 Oct;51(5):2256-2267. doi: 10.3758/s13428-018-1152-2. PMID 30367386
- [Background] Raven J, Raven J, Court R. Mill Hill Vocabulary Scale. Oxford: Oxford University Press. 1998.
- [Background] Shipley WC. Shipley Institute of Living Scale. Los Angeles, CA: Western Psychological Services. 1986.
- [Background] Rammstedt B, John OP. Measuring personality in one minute or less: A 10-item short version of the Big Five Inventory in English and German. Journal of Research in Personality. 2007; 41: 203-212.
- [Background] Adams J, Priest RF, Prince HT. Achievement motive: Analyzing the validity of the WOFO. Psychology of Women Quarterly. 1985; 9: 357-369.
- [Background] Duckworth AL, Peterson C, Matthews MD, Kelly DR. Grit: perseverance and passion for long-term goals. J Pers Soc Psychol. 2007 Jun;92(6):1087-101. doi: 10.1037/0022-3514.92.6.1087. PMID 17547490
- [Background] Poythress NG, Skeem JL, Weir J, Lilienfeld SO, Douglas KS, Edens JF, Kennealy PJ. Psychometric Properties of Carver and White's (1994) BIS/BAS Scales in a Large Sample of Offenders. Pers Individ Dif. 2008 Dec;45(8):732-737. doi: 10.1016/j.paid.2008.07.021. PMID 19956339
- [Background] Dweck CS. Self-theories and goals: their role in motivation, personality, and development. Nebr Symp Motiv. 1990;38:199-235. No abstract available. PMID 2130257
- [Background] Gong X, Paulson SE. Validation of the Schutte Self-Report Emotional Intelligence Scale With American College Students. Journal of Psychoeducational Assessment. 2018; 36: 175-181.
- [Background] Fleming SM, Lau HC. How to measure metacognition. Front Hum Neurosci. 2014 Jul 15;8:443. doi: 10.3389/fnhum.2014.00443. eCollection 2014. PMID 25076880
- [Background] Stepankova H, Lukavsky J, Buschkuehl M, Kopecek M, Ripova D, Jaeggi SM. The malleability of working memory and visuospatial skills: a randomized controlled study in older adults. Dev Psychol. 2014 Apr;50(4):1049-1059. doi: 10.1037/a0034913. Epub 2013 Nov 11. PMID 24219314
- [Background] Jaeggi SM, Buschkuehl M, Parlett-Pelleriti CM, Moon SM, Evans M, Kritzmacher A, Reuter-Lorenz PA, Shah P, Jonides J. Investigating the Effects of Spacing on Working Memory Training Outcome: A Randomized, Controlled, Multisite Trial in Older Adults. J Gerontol B Psychol Sci Soc Sci. 2020 Jun 2;75(6):1181-1192. doi: 10.1093/geronb/gbz090. PMID 31353413
- [Background] Tsai N, Buschkuehl M, Kamarsu S, Shah P, Jonides J, Jaeggi SM. (Un)Great Expectations: The Role of Placebo Effects in Cognitive Training. J Appl Res Mem Cogn. 2018 Dec;7(4):564-573. doi: 10.1016/j.jarmac.2018.06.001. Epub 2018 Aug 3. PMID 31660288
- [Background] Jaeggi SM, Buschkuehl M, Shah P, Jonides J. The role of individual differences in cognitive training and transfer. Mem Cognit. 2014 Apr;42(3):464-80. doi: 10.3758/s13421-013-0364-z. PMID 24081919
- [Background] Szmalec A, Verbruggen F, Vandierendonck A, Kemps E. Control of interference during working memory updating. J Exp Psychol Hum Percept Perform. 2011 Feb;37(1):137-51. doi: 10.1037/a0020365. PMID 20731517
- [Background] Rubin M. The Perceived Awareness of the Research Hypothesis Scale: Assessing the influence of demand characteristics. 2016. doi: 10.6084/m9.figshare.4315778
- [Background] Rabipour S, Davidson PSR. Do you believe in brain training? A questionnaire about expectations of computerised cognitive training. Behav Brain Res. 2015 Dec 15;295:64-70. doi: 10.1016/j.bbr.2015.01.002. Epub 2015 Jan 12. PMID 25591472

RESULTS

PARTICIPANT FLOW:
Groups:
- True Cognitive Training Placebo (Young Adult); True Cognitive Training Placebo (Older Adult): Participants will receive a positive expectation message (e.g., "Previous research has shown that training with this program improves performance on other tasks.") and will complete approximately 7 hours of a cognitive training program that has previously been shown to improve cognition.
  True Cognitive Training Program: The training program is a personal device-based adaptive version of a visual N-back task.
  Positive Expectation Induction: The message given to the participants emphasizes that the given training results in a positive change in cognitive abilities.
- True Cognitive Training Nocebo (Young Adult); True Cognitive Training Nocebo (Older Adult): Participants will receive a negative expectation message (e.g., "Previous research has shown that training with this program decreases performance on other tasks.") and will complete approximately 7 hours of a cognitive training program that has previously been shown to improve cognition.
  True Cognitive Training Program: The training program is a personal device-based adaptive version of a visual N-back task.
  Negative Expectation Induction: The message given to the participants emphasizes that the given training results in a negative change in cognitive abilities.
- Control Cognitive Training Placebo (Young Adult): Participants will receive a positive expectation message (e.g., "Previous research has shown that training with this program increases performance on other tasks.") and will complete approximately 7 hours of control training program that has not previously been shown to improve cognition.
  Control Cognitive Training Program: The training program is a personal device-based adaptive version of a knowledge task (control).
  Positive Expectation Induction: The message given to the participants emphasizes that the given training results in a positive change in cognitive abilities.
- Control Cognitive Training Nocebo (Young Adult): Participants will receive a negative expectation message (e.g., "Previous research has shown that training with this program decreases performance on other tasks.") and will complete approximately 7 hours of control training program that has not previously been shown to improve cognition.
  Control Cognitive Training Program: The training program is a personal device-based adaptive version of a knowledge task (control).
  Negative Expectation Induction: The message given to the participants emphasizes that the given training results in a negative change in cognitive abilities.
Period: Overall Study
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
Started | 66 | 68 | 66 | 63 | 12 | 12
Completed | 45 | 49 | 50 | 49 | 9 | 11
Not Completed | 21 | 19 | 16 | 14 | 3 | 1

BASELINE CHARACTERISTICS:
Population: 28 participants were excluded due to clear noncompliance with the training directions (e.g., did not complete training sessions on time, completed too many).13 participants had missing data due to computer errors on at least 1 task, and 27 participants scored outside of 3 standard deviations from the mean on at least 1 task and were also excluded from all analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult) | Total
Number analyzed (Participants) | 30 | 32 | 36 | 27 | 9 | 11 | 145
Age, Continuous [Mean (Standard Deviation); unit: years]
  Overall Age | 20.13 (2.58) | 19.59 (1.43) | 20.17 (2.05) | 20.93 (4.88) | 73.11 (6.43) | 70.45 (4.55) | 27.33 (18.18)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 10 | 7 | 9 | 5 | 4 | 1 | 36
  Female | 20 | 25 | 26 | 21 | 5 | 10 | 107
  Non-Binary | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Did not report | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 7 | 4 | 1 | 1 | 29
  Not Hispanic or Latino | 22 | 24 | 28 | 23 | 8 | 9 | 114
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 14 | 16 | 16 | 16 | 0 | 1 | 63
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1 | 0 | 2
  White | 11 | 9 | 11 | 7 | 8 | 10 | 56
  More than one race | 2 | 4 | 4 | 2 | 0 | 0 | 12
  Unknown or Not Reported | 2 | 3 | 5 | 2 | 0 | 0 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 32 | 36 | 27 | 9 | 11 | 145
n-back baseline performance [Mean (Standard Deviation); unit: score on a scale] | .58 (.19) | .52 (.19) | .59 (.20) | .58 (.17) | .52 (.17) | .50 (.11) | .57 (.19)
O-span baseline performance [Mean (Standard Deviation); unit: Letter sets correctly recalled] | 42.87 (18.51) | 43.97 (17.90) | 38.81 (14.94) | 36.93 (19.53) | 11.13 (8.20) | 16.09 (10.31) | 37.17 (19.06)
Task-Switching Task baseline performance [Mean (Standard Deviation); unit: milliseconds] | 588.27 (321.44) | 535.21 (286.86) | 585.39 (264.37) | 630.44 (292.10) | 406.56 (215.71) | 511.65 (356.46) | 566.61 (292.11)
Countermanding baseline performance [Mean (Standard Deviation); unit: milliseconds] | 56.50 (57.32) | 50.66 (68.93) | 61.72 (66.27) | 56.62 (66.48) | 25.20 (64.48) | 67.35 (90.92) | 55.62 (66.59)
UFOV baseline performance [Mean (Standard Deviation); unit: milliseconds] | 63.18 (19.47) | 55.35 (13.77) | 61.08 (16.02) | 61.87 (24.49) | 122.48 (39.62) | 162.12 (44.34) | 71.52 (37.41)
ANT baseline performance [Mean (Standard Deviation); unit: milliseconds] | 91.93 (54.52) | 96.54 (43.61) | 99.47 (37.52) | 90.03 (59.28) | 132.06 (53.48) | 89.93 (50.59) | 96.81 (49.17)
Mental Rotation baseline performance [Mean (Standard Deviation); unit: proportion correct] | .68 (.19) | .73 (.19) | .75 (.17) | .76 (.16) | .79 (.21) | .62 (.15) | .72 (.18)
Paper Folding baseline performance [Mean (Standard Deviation); unit: proportion correct] | .67 (.17) | .67 (.18) | .64 (.22) | .70 (.20) | .44 (.21) | .26 (.09) | .63 (.22)
RAPM baseline performance [Mean (Standard Deviation); unit: proportion correct] | .58 (.17) | .55 (.19) | .62 (.20) | .60 (.23) | .48 (.17) | .29 (.13) | .56 (.21)
UCMRT baseline performance [Mean (Standard Deviation); unit: proportion correct] | .68 (.15) | .60 (.19) | .63 (.19) | .62 (.21) | .34 (.13) | .36 (.17) | .59 (.21)
Mill Hill vocabulary baseline performance [Mean (Standard Deviation); unit: proportion correct] | .58 (.12) | .56 (.17) | .57 (.11) | .56 (.11) | .69 (.16) | .69 (.07) | .59 (.13)
Shipley vocabulary baseline performance [Mean (Standard Deviation); unit: proportion correct] | .75 (.10) | .75 (.14) | .84 (.12) | .82 (.12) | .84 (.16) | .85 (.11) | .81 (.13)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Correct Targets Identified Minus False Identifications in the n-Back Task
Description: The n-Back Task is a measure of working memory. The participant is sequentially shown a series of letters and is asked to indicate whether the current letter matches the letter presented "n" items before. The n levels range between 1- and 3-back. Each level of n-back has 17-19 letters, with 5 target letters. The dependent measure is the proportion of correctly identified targets minus the proportion of incorrectly identified non-targets. Scores range from 0-1. Higher scores indicate better performance.
Time Frame: post-test 1 at 25 days, post-test 2 at 34 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
Number analyzed (Participants) | 30 | 32 | 36 | 27 | 9 | 11
score on a scale
  Post-test 1 | .80 (.20) | .70 (.22) | .68 (.22) | .21 (.19) | .70 (.08) | .69 (.19)
  Post-test 2 | .80 (.23) | .73 (.21) | .68 (.23) | .60 (.35) | .71 (.12) | .71 (.13)

2. Primary Outcome: Number of Correctly Recalled Letter Sets in the O-Span Task
Description: The O-Span Task is a measure of working memory. In each trial, the participant is alternately presented with a simple math equation and a letter and then is asked to recall the sequence of letters in order. The participant will complete 15 trials, which vary between 3-7 math problem/letter pairs. The dependent measure is the total number of letters in correctly recalled trials. Scores range from 0 to 75. Higher scores indicate better performance.
Time Frame: post-test 1 at 25 days, post-test 2 at 34 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
Number analyzed (Participants) | 30 | 32 | 36 | 27 | 9 | 11
score on a scale
  Post-test 1 | 47.07 (18.79) | 43.07 (21.11) | 41.78 (18.21) | 43 (23.03) | 20.22 (11.51) | 19.72 (10.76)
  Post-test 2 | 42.2 (19.11) | 43.56 (20.57) | 42.61 (19.92) | 38.85 (23.49) | 20.11 (9.20) | 21.72 (11.15)

3. Primary Outcome: Difference in Response Time Between Switch Trials and Non-switch Trials (Switch Cost) in the Task Switching Task
Description: The Task Switching task is a measure of cognitive flexibility. On each trial, participants view a letter and a digit. The location of the pair instructs the participants to either categorize the letter as a consonant or vowel or else categorize the digit as even or odd. Trials can be either "non-switch trials" - in which the participant is asked to perform the same task as on the previous trial - or "switch trials" - in which the participant is asked to perform the opposite task as on the previous trial. The participant will complete 48 trials. A "switch cost" is calculated by subtracting the average response time for non-switch trials from the average response time for switch trials (milliseconds). Lower scores indicate better performance.
Time Frame: post-test 1 at 25 days, post-test 2 at 34 days
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
Number analyzed (Participants) | 30 | 32 | 36 | 27 | 9 | 11
milliseconds
  Post-test 1 | 435.79 (274.42) | 471.14 (240.36) | 384.51 (186.88) | 529.88 (318.02) | 503.74 (292.83) | 529.42 (372.15)
  Post-test 2 | 388.21 (186.16) | 441.86 (310.86) | 347.63 (193.71) | 506.94 (349.17) | 519.73 (234.29) | 519.05 (208.95)

4. Primary Outcome: Difference in Response Time Between Switch Trials and Non-switch Trials (Switch Cost) in the Countermanding Task
Description: The Countermanding task is a measure of cognitive flexibility. Participants are presented with two types of stimuli on either the right or the left side of the screen and are required to tap on one of two buttons on either the same side as the stimulus or on the opposite side of the stimulus. Trials can be either "non-switch trials" - in which the participant is asked to perform the same task as on the previous trial - or "switch trials" - in which the participant is asked to perform the opposite task as on the previous trial. The participant will complete 48 trials. A switch cost is calculated by subtracting the average response time for non-switch trials from the average response time for switch trials (in milliseconds). Lower scores indicate better performance.
Time Frame: post-test 1 at 25 days, post-test 2 at 34 days
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
Number analyzed (Participants) | 30 | 32 | 36 | 27 | 9 | 11
milliseconds
  Post-test 1 | 67.89 (51.71) | 51.89 (57.14) | 47.48 (56.06) | 39.67 (62.96) | 32.53 (81.26) | -11.46 (138.73)
  Post-test 2 | 52.92 (85.02) | 31.27 (57.47) | 33.90 (74.61) | 46.56 (57.17) | 23.19 (63.25) | -3.92 (53.12)

5. Primary Outcome: Threshold of Response Time in the Useful Field of View (UFOV) Task
Description: The UFOV is a measure of visual selective attention. Participants are briefly presented with a display consisting of 24 items (3 on each of the four radial spokes and the four obliques; evenly spaced). One of the items is a target, while the remaining items are distractors. The participants' task is to indicate upon which of the 8 spokes the target appeared. The display times vary between 16-500ms. The task uses an adaptive staircase procedure, in which the display times increase or decrease based on the participant's performance, to calculate the participant's response threshold in milliseconds. Lower threshold scores indicate better performance
Time Frame: post-test 1 at 25 days, post-test 2 at 34 days
Measure: Median (Standard Deviation); unit: milliseconds
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
Number analyzed (Participants) | 30 | 32 | 36 | 27 | 9 | 11
milliseconds
  Post-test 1 | 52.60 (14.82) | 50.46 (16.78) | 52.18 (16.30) | 56.71 (23.70) | 123.05 (21.46) | 137.21 (46.19)
  Post-test 2 | 49.66 (17.02) | 49.11 (14.59) | 47.89 (14.49) | 53.81 (21.33) | 119.34 (30.49) | 141.92 (49.94)

6. Primary Outcome: Difference in Response Time of Compatible Trials and Incompatible Trials in the Attentional Network Task (ANT)
Description: The ANT is a measure of visual selective attention. On each trial, participants view a center arrow that faces either left or right. The arrow can be flanked on either side by either response compatible arrows (i.e., arrows facing in the same direction as the center arrow) or response incompatible arrows (i.e., facing the other direction). The participants' task is to indicate the direction that the center arrow is pointing. Participants will complete 96 trials. The compatibility effect is calculated by subtracting the average response time of compatible trials from the average response time of incompatible trials (in milliseconds). Lower scores indicate better performance.
Time Frame: post-test 1 at 25 days, post-test 2 at 34 days
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
Number analyzed (Participants) | 30 | 32 | 36 | 27 | 9 | 11
milliseconds
  Post-test 1 | 90.67 (37.65) | 92.12 (60.67) | 90.52 (39.05) | 98.44 (49.15) | 88.66 (32.16) | 80.33 (52.28)
  Post-test 2 | 84.60 (44.95) | 86.55 (45.55) | 82.10 (32.01) | 89.22 (46.20) | 70.25 (39.10) | 113.69 (30.74)

7. Primary Outcome: Proportion of Correct Responses on the Mental Rotation Task
Description: The mental rotation task is a measure of spatial cognition. Each trial displays two 2-D images, and the participant is asked whether the image on the right is a rotated version or a mirror-reserved and rotated version of the image on the left. The participant will complete 36 trials.
Time Frame: post-test 1 at 25 days, post-test 2 at 34 days
Measure: Mean (Standard Deviation); unit: proportion correct
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
Number analyzed (Participants) | 30 | 32 | 36 | 27 | 9 | 11
proportion correct
  Post-test 1 | .77 (.18) | .81 (.18) | .81 (.16) | .81 (.16) | .82 (.19) | .74 (.13)
  Post-test 2 | .80 (.18) | .82 (.18) | .82 (.18) | .84 (.16) | .80 (.20) | .80 (.15)

8. Primary Outcome: Proportion of Correct Responses in the Paper Folding Task
Description: The Paper Folding task is a measure of mental rotation. Participants are shown 2-4 images depicting a piece of paper being folded with a hole being punched after the last fold. The participant is asked to imagine and indicate what the paper would look like unfolded. The participant will complete 10 trials.
Time Frame: post-test 1 at 25 days, post-test 2 at 34 days
Measure: Mean (Standard Deviation); unit: proportion correct
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
Number analyzed (Participants) | 30 | 32 | 36 | 27 | 9 | 11
proportion correct
  Post-test 1 | .74 (.21) | .73 (.18) | .72 (.18) | .66 (.22) | .46 (.17) | .36 (.15)
  Post-test 2 | .76 (.17) | .76 (.17) | .74 (.21) | .73 (.23) | .45 (.18) | .42 (.13)

9. Primary Outcome: Proportion of Correct Responses in Raven's Advanced Progressive Matrices Task
Description: Raven's Advanced Progressive Matrices task is a measure of fluid intelligence. The participant is presented with a grid of elements with one of the elements missing and is asked to identify the missing element that completes the grid pattern. The participant will complete 14 trials.
Time Frame: post-test 1 at 25 days, post-test 2 at 34 days
Measure: Mean (Standard Deviation); unit: proportion correct
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
Number analyzed (Participants) | 30 | 32 | 36 | 27 | 9 | 11
proportion correct
  Post-test 1 | .67 (.18) | .58 (.19) | .65 (.17) | .54 (.19) | .42 (.17) | .36 (.16)
  Post- test 2 | .66 (.18) | .61 (.20) | .68 (.21) | .65 (.20) | .33 (.19) | .33 (.10)

10. Primary Outcome: Proportion of Correct Responses in the UC Matrix Reasoning Task
Description: The UC Matrix Reasoning task is a measure of fluid intelligence. The participant is presented with a grid of elements with one of the elements missing and is asked to identify the missing element that completes the grid pattern. The participant will complete 16 trials.
Time Frame: post-test 1 at 25 days, post-test 2 at 34 days
Measure: Mean (Standard Deviation); unit: proportion correct
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
Number analyzed (Participants) | 30 | 32 | 36 | 27 | 9 | 11
proportion correct
  Post-test 1 | .74 (.14) | .69 (.20) | .73 (.17) | .67 (.22) | .44 (.18) | .39 (.22)
  Post-test 2 | .75 (.18) | .70 (.19) | .74 (.18) | .90 (.21) | .42 (.12) | .42 (.14)

11. Primary Outcome: Proportion of Correct Responses in the Mill-Hill Vocabulary Scale
Description: In this vocabulary task, participants are asked to select the appropriate synonym for a target word among several alternatives for 25 words.
Time Frame: post-test 1 at 25 days, post-test 2 at 34 days
Measure: Mean (Standard Deviation); unit: proportion correct
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
Number analyzed (Participants) | 30 | 32 | 36 | 27 | 9 | 11
proportion correct
  Post-test 1 | .58 (.15) | .59 (.18) | .58 (.14) | .59 (.11) | .66 (.16) | .70 (.10)
  Post-test 2 | .58 (.13) | .61 (.17) | .61 (.12) | .59 (.14) | .65 (.13) | .70 (.08)

12. Primary Outcome: Proportion of Correct Responses in the Shipley Institute of Living Scale
Description: Participants will complete Part I of the Shipley Institute of Living Scale, which is a measure of vocabulary. Participants are asked to select the appropriate synonym for a target word among several alternatives for 15 words.
Time Frame: post-test 1 at 25 days, post-test 2 at 34 days
Measure: Mean (Standard Deviation); unit: proportion correct
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
Number analyzed (Participants) | 30 | 32 | 36 | 27 | 9 | 11
proportion correct
  Post-test 1 | .80 (.12) | .79 (.13) | .77 (.10) | .77 (.10) | .86 (.01) | .91 (.07)
  Post-test 2 | .77 (.11) | .77 (.15) | .84 (.11) | .81 (.14) | .89 (.09) | .90 (.11)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 34 days
Description: This study posed no adverse risks.
Arm/Group | True Cognitive Training Placebo (Young Adult) | True Cognitive Training Nocebo (Young Adult) | Control Cognitive Training Placebo (Young Adult) | Control Cognitive Training Nocebo (Young Adult) | True Cognitive Training Placebo (Older Adult) | True Cognitive Training Nocebo (Older Adult)
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/68 | 0/66 | 0/63 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/68 | 0/66 | 0/63 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/66 | 0/68 | 0/66 | 0/63 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT04344028/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT04344028/ICF_001.pdf